CLINICAL TRIAL: NCT05191992
Title: Basic Life Support (BLS) Training by Homemade Manikin in Undergraduate Nursing Students
Brief Title: Basic Life Support (BLS) Training by Homemade Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Nurten Taşdemir (Unknown)
Responsible Party: Principal Investigator, Dilek YILDIRIM TANK, PhD. Research Assistant, Zonguldak Bulent Ecevit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CPRhandmade
Record Dates: First submitted 2021-11-16; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation; Education, Nursing
Keywords: nursing student; cardiopulmonary resuscitation; mannequins; education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): The group will receive CPR training with the e-learning method and will learn skills with a handmade mannequin.
  Interventions: Other: CPR training with e-learning with a handmade mannequin.

INTERVENTIONS:
Other: CPR training with e-learning with a handmade mannequin. — The group, who was given theory training with the e learning method, will be taught to make pillows and plastic bottles and cpr mannequins, and they will be asked to practice. Knowledge and skills assessment will be made before, immediately after and 1 month after the training.

SUMMARY:
The experimentally planned research was carried out between the dates of 01.06.2021-10.11.2021 with the students of ……………. Faculty of Health Sciences, Department of Nursing. The students, whose informed consent form was obtained beforehand, were provided to fill in the Participant Diagnosis Form and the Basic Life Support Information Evaluation Form questioning their demographic characteristics before the education. Afterward, with the e-learning method (Perculus 3 Virtual Classroom), the students have given Basic Life Support training in accordance with the AHA 2020 guidelines through a Powerpoint presentation. After the training, the information evaluation form was filled in again by the students in an electronic environment. Afterward, the students were shown how to make a Basic Life Support manikin with a pillow and plastic pet bottle, and the CPR performance was explained with the manikin. The students who made the performance in the home environment made a video recording and uploaded the videos they took to the system within 1 day. Two researchers who are experts in their fields made the video evaluations according to the basic life support performance evaluation form. Later, in the online debriefing session, the pros and cons of the training were discussed with the students, and after 1 month, knowledge and skills were evaluated again and the level of permanence on the subject was measured.

DETAILED DESCRIPTION:
Cardiovascular diseases are in the first place among the causes of death, causing 31% (17.9 million) of all deaths worldwide. Considering deaths worldwide, 200,000 people can be revived each year with early cardiopulmonary resuscitation (CPR) and effective care thereafter.

The International Liaison Committee on Resuscitation defines Basic Life Support (BLS) as "providing adequate circulation and respiration until advanced life support conditions are met to save lives and prevent worsening of the patient's condition in case of cardiopulmonary arrest. The critical period after the cessation of cardiac and respiratory function, in which vital signs disappear but the loss is reversible, is the subject of BLS. After sudden cardiac arrest, brain cells can only withstand oxygen deprivation for 3-5 minutes, so when BLS practice is started within the first four minutes, the survival rate is 29%, while when started after the first four minutes, the survival rate drops to 7%. Few of the patients who are revived after four minutes are able to maintain their previous quality of life. Effective implementation of this practice, which significantly reduces mortality and morbidity, is very important.

It is very important that the knowledge and skills of the students of the nursing department, who have a high probability of encountering first aid applications due to their professional life and are expected to perform these applications correctly, are sufficient and up-to-date. As a reflection of this, First Aid and Emergency Care Nursing course have taken its place in the curriculum as a compulsory vocational course within the scope of the Nursing National Core Education Program in higher education institutions providing nursing education, and it has been provided to be carried out theoretically and practically.

The quality of cardiopulmonary resuscitation includes providing adequate chest compressions, providing adequate depth of chest compressions, allowing chest reinstatement between compressions, minimizing interruptions in chest compressions, and avoiding excessive ventilation. Cardiopulmonary resuscitation training is carried out in laboratory environments, especially with cardiopulmonary resuscitation manikins. However, the difficulty of accessing these manikins and their high cost are especially important in recent days. The necessity brought by the recent pandemic process, or the difficulty of accessing manikins that require high resources in educational environments where the transition to e-learning is attempted, causes an increase in the knowledge and skills gap that already exists in this regard. Studies have reported that the effectiveness of BLS training decreases over time. It is expected that the education method supported by e-learning and accessible materials will contribute to the permanence of education by allowing the application to be repeated independently of time, place, and expensive materials.

Homemade manikins developed with low-cost limited materials for CPR training began to be discovered many years ago but were not widely used. This study was conducted in order to measure the effectiveness and permanence of the CPR training given with homemade manikins in this period when e-learning became widespread.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate the study,
* Having taken basic nursing education courses

Exclusion Criteria:

* Not wanting to participate in the study,
* Not taking basic nursing education courses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Increasing the effectiveness of BLS training on knowledge given with by e-learning method | 1 month
  CPR training given with the e-learning method cannot contribute to skill development since there is no mannequin access. The opportunity to practice with the handmade, inexpensive mannequin provided ensures that the training is effective. The effectiveness of the training was evaluated with the 10-question BLS knowledge evaluation form which was organized according to the AHA guideline by authors. In the evaluation of the 10-question knowledge test, each question is 1 point. If the evaluation score is over 70%, it indicates that the participant is successful.
Increasing the effectiveness of BLS training on skills given with by e-learning method | 1 month
  CPR training given with the e-learning method cannot contribute to skill development since there is no mannequin access. The opportunity to practice with the handmade, inexpensive mannequin provided ensures that the training is effective. The effectiveness of the training was evaluated with the 20-item BLS Skills Assessment Form, which was organized according to the AHA guideline by authors. In the evaluation of the 20-question BLS Skills Assessment Form, each item is 1 point. If the assessment score is over 70%, it indicates that the participant is successful.
Increasing the permanence of BLS training on knowledge given by e-learning method | 1 month
  Studies have reported that the effectiveness of BLS training decreases over time. It is expected that the education method supported by e-learning and handmade mannequins will contribute to the permanence of education by allowing the application to be repeated independently of time, place, and expensive materials. The permanence of the training was evaluated with the 10-question BLS knowledge evaluation form which was organized according to the AHA guideline by authors. In the evaluation of the 10-question knowledge test, each question is 1 point. If the evaluation score is over 70%, it indicates that the participant is successful.
Increasing the permanence of BLS training on skills given by e-learning method | 1 month
  Studies have reported that the effectiveness of BLS training decreases over time. It is expected that the education method supported by e-learning and handmade mannequins will contribute to the permanence of education by allowing the application to be repeated independently of time, place, and expensive materials. The permanence of the training was evaluated with the 20-item BLS Skills Assessment Form, which was organized according to the AHA guideline by authors.
  In the evaluation of the 20-question BLS Skills Assessment Form, each item is 1 point. If the assessment score is over 70%, it indicates that the participant is successful.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months

REFERENCES:
- See also: Basic Life Support: an accessible tool in layperson training — http://dx.doi.org/10.1590/1806-9282.65.10.1300